CLINICAL TRIAL: NCT00917319
Title: Randomized Controlled Study on Effectiveness of Implementing Bundling Infection Control Interventions for Prevention and Control of Healthcare-Associated Infections in General Medical Wards at Siriraj Hospital, Bangkok, Thailand
Brief Title: Prevention and Control of Healthcare-Associated Infections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Visanu Thamlikitkul, Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Siriraj CEU 52-001; Siriraj Hospital
Record Dates: First submitted 2009-06-05; First posted 2009-06-10 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Nosocomial Infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infection control measure (Experimental): Bundling Infection Control Interventions
  Interventions: Other: Bundling Infection Control Interventions

INTERVENTIONS:
Other: Bundling Infection Control Interventions — identify risk factors for developing HAIs, receive general infection control measures as well as infection control measures appropriate for the identified risk factor (s)

SUMMARY:
Bundling infection control interventions should decrease incidence of Healthcare-Associated Infections in General Medical Wards at Siriraj Hospital, Bangkok, Thailand

ELIGIBILITY:
Inclusion Criteria:

* The patients hospitalized to general medical wards

Exclusion Criteria:

* The patients hospitalized less than 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of healthcare-associated infection | 7 months

SECONDARY OUTCOMES:
Incidence of hospital-acquired pneumonia and catheter-associated UTI | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Visanu Thamlikitkul, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Department of Medicine, Faculty of Medicine Siriraj Hospital, Bangkoknoi,, Bangkok, Thailand

REFERENCES:
- [Derived] Korbkitjaroen M, Vaithayapichet S, Kachintorn K, Jintanothaitavorn D, Wiruchkul N, Thamlikitkul V. Effectiveness of comprehensive implementation of individualized bundling infection control measures for prevention of health care-associated infections in general medical wards. Am J Infect Control. 2011 Aug;39(6):471-6. doi: 10.1016/j.ajic.2010.09.017. Epub 2011 May 12. PMID 21565423